CLINICAL TRIAL: NCT01003964
Title: Randomized phase2 Study of IP vs. GP as the First-line Therapy Followed by Two Different Sequences as the 2nd or 3rd-line Therapy for Patients With Advanced NSCLC;
Brief Title: Pharmacogenomic Study for Providing Personalized Strategy to the Treatment of Non-small Cell Lung Cancer (NSCLC) IIIB/IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-08-371
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NON-SMALL CELL LUNG CANCER; excision repair cross-complementing 1; Gemcitabine and cisplatin; Irinotecan and cisplatin; advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GP group (Experimental): Gemcitabine (1250 mg/m2) IV on D 1, 8. Cisplatin (75 mg/m2) IV on D1 every 3 weeks.
  Interventions: Drug: GP
- IP group (Experimental): Irinotecan (65 mg/m2) IV on day1 , 8 Cisplatin (30 mg/m2) IV on day 1 , 8 every 3 weeks
  Interventions: Drug: IP

INTERVENTIONS:
Drug: IP — Irinotecan (65 mg/m2) IV on day1 , 8 Cisplatin (30 mg/m2) IV on day 1 , 8 every 3 weeks
  Other Names: Irrinotecan, Cisplatin
  Arms: IP group
Drug: GP — Gemcitabine (1250 mg/m2) IV on D 1, 8. Cisplatin (75 mg/m2) IV on D1 every 3 weeks.
  Other Names: Gemcitabine, Cisplatin
  Arms: GP group

SUMMARY:
The primary objective of this randomized phase II study is to compare the Response Rate of each sequence of treatment approach in patients with advanced NSCLC. Additionally, development of gene expression profiles and genotypes that can predict response to commonly used chemotherapy may provide a unique opportunity to better utilize drugs shown to be effective in first- or second-line therapy. Here, the investigators will conduct a pharmacogenomic study to provide rational approach to the treatment of NSCLC by developing predictors of cisplatin (first-line agent) and pemetrexed or docetaxel (second-line agents) sensitivity and demonstrating the clinical value of identifying the most appropriate drug on the basis of sensitivity profile for the treatment regimen of each individual patient. Such an approach is likely to maximize response to chemotherapy and may change the current empirical paradigm of NSCLC therapy.

DETAILED DESCRIPTION:
Cisplatin-based chemotherapy is currently considered to be the standard treatment in advanced non-small cell lung cancer (NSCLC). However, overall response is only 30-40%, suggesting that a majority of the patients do not respond to platinum. Subsequently, those patients who experience treatment failure with platinum-based therapy typically received pemetrexed or docetaxel as second-line treatment, with response rate of approximately 7% to 10%. The primary objective of this randomized phase II study is to compare the Response Rate of each sequence of treatment approach in patients with advanced NSCLC. Additionally, development of gene expression profiles and genotypes that can predict response to commonly used chemotherapy may provide a unique opportunity to better utilize drugs shown to be effective in first- or second-line therapy. Here, we will conduct a pharmacogenomic study to provide rational approach to the treatment of NSCLC by developing predictors of cisplatin (first-line agent) and pemetrexed or docetaxel (second-line agents) sensitivity and demonstrating the clinical value of identifying the most appropriate drug on the basis of sensitivity profile for the treatment regimen of each individual patient. Such an approach is likely to maximize response to chemotherapy and may change the current empirical paradigm of NSCLC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of NSCLC, Stage IV or selected stage IIIB (malignant pleural or pericardial effusion or supraclavicular adenopathy) according to the American Joint Committee on Cancer (AJCC).
* Adequate tumor tissues for ERCC1 analysis.
* No prior chemotherapy.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
* No other forms of cancer therapy, such as radiation, immunotherapy and major surgery for at least 3 weeks before the enrollment in study.
* Performance status of 0, 1, or 2 on the ECOG criteria.
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumors(RECIST), the presence of at least one unidimensionally measurable lesion with longest diameter 10mm by spiral CT scan.
* Estimated life expectancy of at least 12 weeks.
* Patient compliance that allow adequate follow-up.
* Adequate hematologic and renal function.
* Informed consent from patient or patient's relative.
* Males or females at least 18 years of age.
* No pregnancy or breast feeding.
* Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs

Exclusion Criteria:

* MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia.
* Serious concomitant infection.
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2009-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response Rate | every 6 weeks

SECONDARY OUTCOMES:
Overall survival (OS) | every 8 weeks
  from the first day of treatment to death
Progression-free survival (PFS) | every 6 weeeks
  as the period between the day of the treatment and the date of progression or death
adverse event | every 3 weeks
  from C1D1 to 30 days after the last dose administration
Pharmacogenomic study using tumor tissue and blood for providing rational strategy to the treatment of advanced NSCLC | 2 times
  at baseline and time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: JI-YOUN HAN, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JY, Choi JJ, Kim JY, Han YL, Lee GK. PNA clamping-assisted fluorescence melting curve analysis for detecting EGFR and KRAS mutations in the circulating tumor DNA of patients with advanced non-small cell lung cancer. BMC Cancer. 2016 Aug 12;16:627. doi: 10.1186/s12885-016-2678-2. PMID 27519791